CLINICAL TRIAL: NCT04556071
Title: A Single-arm, Prospective, Open-label, Phase II Study to Evaluate the Efficacy and Safety of Niraparib Combined With Bevacizumab in Platinum Refractory/Resistant Recurrent Ovarian, Fallopian Tube or Peritoneal Cancer
Brief Title: Efficacy and Safety of Niraparib Combined With Bevacizumab in Platinum Refractory/Resistant Recurrent Ovarian Cancer
Acronym: AVANIRA3
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiaoxiang Chen (Other)
Responsible Party: Sponsor-Investigator, Xiaoxiang Chen, Academic secretary of gynecological oncology Committee of Jiangsu anti cancer association, Jiangsu Cancer Institute & Hospital
Organization: Jiangsu Cancer Institute & Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JiangsuCH001
Record Dates: First submitted 2020-09-15; First posted 2020-09-21 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Ovarian Neoplasms; Fallopian Tube Neoplasms; Endocrine Gland Neoplasms; Neoplasms by Site; Neoplasms; Genital Neoplasms, Female; Urogenital Neoplasms; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Carcinoma, Ovarian Epithelial; Ovarian Diseases; Adnexal Diseases; Genital Diseases, Female; Endocrine System Diseases; Gonadal Disorders; Carcinoma; Bevacizumab; Enzyme Inhibitors; Antineoplastic Agents; Molecular Mechanisms of Pharmacological Action; Angiogenesis; BRCA1 Mutation; BRCA2 Mutation; Homologous Recombination Deficiency
Keywords: Platinum Refractory/Resistant Recurrent Ovarian Cancer; Niraparib; Bevacizumab; homologous recombination deficiency; tumor burden
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Endocrine Gland Neoplasms; Neoplasms by Site; Neoplasms; Genital Neoplasms, Female; Urogenital Neoplasms; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Carcinoma, Ovarian Epithelial; Ovarian Diseases; Adnexal Diseases; Genital Diseases, Female; Endocrine System Diseases; Gonadal Disorders; Carcinoma | interventions — niraparib; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Niraparib-bevacizumab combination (Experimental): Niraparib-bevacizumab combination therapy until disease progression
  Interventions: Drug: Niraparib; Drug: Bevacizumab

INTERVENTIONS:
Drug: Niraparib — Niraparib will be administered orally once a day continuously throughout each 21-days cycle. The initial dose will be based on the participant's basal body weight or platelet count. Participants with basal body weight≥77 kg and basal platelet count of≥150,000/microliter (μL) will take 300 mg daily. While participants with basal body weight<77 kg and/or basal platelet count <150,000/μL will take 200 mg daily.
  Other Names: Zejula
Drug: Bevacizumab — The dose of Bevacizumab will be 15 mg/kg that administered via a 30-minute intravenous infusion on day 1 of every 21-day cycle in the absence of progressive disease (PD), unacceptable toxicity, participant withdrawal, Investigator's decision, or death.
  Other Names: Avastin

SUMMARY:
Niraparib is an oral, potent and highly selective PARP1/2 inhibitor. It can be used as a single drug in HRD positive ovarian cancer patients for multi-line therapy. Bevacizumab is a recombinant humanized monoclonal antibody that inhibits tumor angiogenesis and is also recommended for the treatment of recurrent ovarian cancer. Clinical studies showed that niraparib combined with bevacizumab could significantly prolong progression free survival of platinum sensitive recurrent ovarian cancer. We intend to conduct a single-arm, prospective, open-label, phase II study to observe the efficacy and safety of niraparib combined with bevacizumab in the treatment of FIGO III/IV platinum refractory/resistant ovarian cancer, fallopian tube cancer and primary peritoneal cancer. The results are expected to provide more effective and precise treatment for platinum resistant recurrent/refractory ovarian cancer patients.

DETAILED DESCRIPTION:
The study is a single-arm, prospective, open-label, phase II study to observe the efficacy and safety of niraparib combined with bevacizumab in the treatment of FIGO III/IV platinum refractory/resistant ovarian cancer, fallopian tube cancer and primary peritoneal cancer.The primary end point is the objective response rate, and the secondary end points are progression free survival, duration of remission, disease control rate and safety. We also stratified analysis the level of tumor load, the status of BRCA and HRD on the efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects understand the trial process, sign informed consent, agree to participate in the study, and have the ability to follow the protocol;
2. Participant must be female ≥18 years of age;
3. Histologically confirmed FIGO stage III or IV ovarian cancer, fallopian tube cancer, or primary peritoneal cancer;
4. Participants must have high-grade serous or endometrioid histology;
5. Subjects were initially treated with platinum, and the disease recurrence occurred within 6 months after the end of the previous platinum-containing chemotherapy, that is, platinum resistance relapsed; Subjects have disease progression during initial platinum based chemotherapy defined as platinum refractory;
6. Patients may have received a PARP inhibitor as first-line maintenance therapy;
7. Patients may have received bevacizumab though no other prior use of anti-angiogenic therapy；
8. Subjects must have measurable lesions (according to RECIST1.1) and radiologically confirmed disease progression at the time of previous treatment; or CA125 elevated for two consecutive times and 2.5 times upper the limit of normal value；
9. Subject agrees to take blood samples for gBRCA mutations, can provide formalin-fixed, paraffin-embedded tumor tissue samples for sBRCA and homologous recombination deficiency(HRD) detection;
10. Life expectancy>12 weeks;
11. Subject's ECOG physical status score is 0-2;
12. Good organ function, including:Neutrophil count≥1500/μL;Platelets≥100,000/μL;Hemoglobin≥10g/dL;Serum creatinine≤1.5 times the upper limit of normal value, or creatinine clearance≥60mL/min (calculated according to Cockcroft-Gault formula);Total bilirubin≤1.5 times the upper limit of normal value or direct bilirubin≤ 1.0 times the upper limit of normal value;AST and ALT≤2.5 times the upper limit of normal value. When liver metastases are present, it must be≤5 times the upper limit of normal value;
13. For women with fertility potential, if blood test or urine pregnancy test is negative within one week before enrollment, effective contraceptive measures must be taken, such as physical barrier contraceptive method (condom) or complete abstinence. Oral, injectable or implantable hormonal contraceptives are not allowed. Or women without reproductive potential, defined as: I. Natural menopause and menopause for more than 1 year; II. Surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy); III. serum follicle-stimulating hormone, luteinizing hormone, and plasma estradiol levels were within the menopausal criteria of the research center laboratory;
14. Subject is able to adhere to the protocol;
15. The adverse effect of any previous chemotherapy have recovered to ≤ Grade1 (CTCAE v5.0) or baseline levels, except for sensory neuropathy or hair loss with stable symptoms ≤ Grade2 (CTCAE v5.0).

Exclusion Criteria:

1. Personnel involved in the formulation or implementation of the research plan;
2. Patient participated in other clinical trails using other experimental drugs at the same time as the study;
3. People who are known to be allergic to Niraparib or Bevacizumab (or active or inactive ingredients of drugs with similar chemical structure);
4. People who are inability to swallow oral drugs and any gastrointestinal diseases that may interfere with the absorption and metabolism of the study drugs, such as uncontrollable nausea and vomiting, gastrointestinal obstruction or malabsorption;
5. Major surgery was performed within 4 weeks before the start of the study or did not recover after the operation;
6. Received palliative radiotherapy of >20% bone marrow 1 week before enrollment;
7. The subjects had other malignant diseases in past 2 years, except skin squamous cell carcinoma, basal-like carcinoma, breast intraductal carcinoma in situ, or cervical carcinoma in situ;
8. Previous or currently diagnosed myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML);
9. Patients with serious and uncontrollable diseases or the general situation of the subjects judged by the researchers to be unsuitable for enrolling the study, including but not limited to: active viral infection, such as human immunodeficiency virus, hepatitis B, hepatitis C, etc.; severe cardiovascular disease, uncontrollable ventricular arrhythmia, myocardial infarction in the last three months; uncontrollable grand mal epilepsy, Unstable spinal cord compression, superior vena cava syndrome or other mental disorders that affect patients to sign the informed consent; hypertension beyond drug control; immune deficiency (except splenectomy) or other diseases that researchers consider may expose patients to high-risk toxicity;
10. The previous history of thromboembolism was defined as: uncontrolled pulmonary embolism, deep venous thrombosis, and other related conditions after anticoagulant therapy for more than 3 months before enrollment;
11. Any medical history or existing clinical evidence indicates that there may be confusion of study results, interference with patients' compliance with the trial protocol throughout the study treatment period, or not in the best interests of patients;
12. Receive platelet or red blood cell transfusions within 4 weeks;
13. Patients who are pregnant or lactation, or who plan to become pregnant during study treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-11-06 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | at 6 months
  ORR is defined as the proportion of participants achieving complete response (CR) or partial response (PR) as assessed by RECIST1.1.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Through study completion, an average of 1 year
  PFS is defined as the time in months from the date of first study drug administration to the date of first documentation of progressive disease (PD) or death as assessed by RECIST1.1.
Disease Control Rate (DCR) | at 6 months
  Disease control rate is defined as the proportion of participants achieving complete response (CR), partial response (PR) or stable disease (SD) according to RECIST1.1.
Duration of Response (DOR) | Through study completion, an average of 1 year
  DOR is defined as the time from the first date of response until the date of first documented progression.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Through study completion, an average of 1 year
  To further describe safety and assess toxicities encountered with the use of the proposed treatment regimen in participants.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoxiang Chen, MD,PhD, Study Chair — Jiangsu Cancer Institute & Hospital
Locations (1):
- JiangSu Cancer Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Contact Prof. Chen for primary data.